CLINICAL TRIAL: NCT06462625
Title: Long-term Clinical and Radiographic Outcomes of Different Knee Osteotomy Techniques for the Treatment of Compartmental Knee Osteoarthritis With Lower Limb Malalignment.
Brief Title: Clinical and Radiological Results of Long Term Tibial and Femoral Osteotomy in Knee Ostheoarthritis With Concomitant Lower Limb Malalignement
Acronym: KNEE OSTEOTOMY
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: KNEE OSTEOTOMY-OA
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis; Malalignment, Bone
MeSH Terms: conditions — Osteoarthritis, Knee; Bone Malalignment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Closing wedge: Patients undergoing closing wedge high tibial osteotomy in knee ostheoarthritis and lower limb malalignement
  Interventions: Other: High tibial osteotomy
- Opening wedge: Patients undergoing opening wedge high tibial osteotomy in knee ostheoarthritis and lower limb malalignement
  Interventions: Other: High tibial osteotomy

INTERVENTIONS:
Other: High tibial osteotomy — Correction of lower limb malalignement with tibial bone wedge insertion/removal

SUMMARY:
The present study aims to evaluate the long-term and medium-term outcomes of different knee osteotomy techniques in the treatment of knee osteoarthritis in patients with lower limb malalignment. This evaluation is necessary in the current context of research on the treatment and prevention of knee osteoarthritis through treatments that do not involve or allow for the postponement of prosthetic replacement. Among the biological treatments performed in orthopedic clinical practice, osteotomy is one of the most promising. However, further long-term evaluations are needed to more clearly determine the indications and potential of this type of intervention, considering the various surgical procedures described for performing it.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing corrective knee osteotomy and any associated procedures such as meniscal repair/resection/replacement, ligament reconstruction, chondral treatment, or regenerative infiltrative treatment;
2. Patients aged between 18 and 70 years at the time of surgical intervention;
3. Patients with isolated compartmental osteoarthritis;
4. Patients with a varus or valgus knee alignment defect of at least 3° compared to mechanical neutrality.

Exclusion Criteria:

1. Patients with advanced multicompartimental osteoarthritis;
2. Patients who are no longer reachable;
3. Women of childbearing age who cannot exclude pregnancy;
4. Patients unable to give informed consent or patients unwilling to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Based on the number of patients treated at Rizzoli with this type of surgical intervention and considering a 25% dropout rate, it is estimated that 150 patients with a follow-up period of 2 to 20 years can be included in the study. It is noteworthy that previous studies with similar aims have a patient sample similar to that proposed by the current study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Score | 24 months after surgery
  It is a validated measurement scale that assesses knee functionality through 8 items, which help determine the condition of the knee in response to the functional demands of daily activities. This evaluation form is commonly used to assess the outcomes of surgery in patients who have undergone operations for ligament or meniscal injuries of the knee. The final score is obtained by summing the various scores from the different items and ranges from 0 to 100. The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) | 24 months after surgery
  The IKDC form is a subjective knee evaluation module that reflects the limitations on activities an individual can perform in daily life and sports, as well as the presence or absence of symptoms. There are three main domains of the IKDC evaluation form: Symptoms, which include pain, stiffness, swelling, and a sense of locking; Sports and daily activities; Current knee function and function before the injury. The questionnaire consists of 10 questions: seven items investigate the patient's symptoms, one item addresses sports participation, one item-comprising 9 points-concerns the difficulties the patient experiences in performing daily activities, and the last item measures the current functionality of the knee.
  The score ranges from 0 to 100, with 100 representing the absence of limitations and symptoms; the further away from this score, the worse the result. The scores can be divided into four groups: excellent (80-100), good (60-80), fair (30-60), and poor (0-30).
Objective IKDC(IKDC standard evaluation form) | 24 months after surgery
  It represents a clinical form completed by the physician following a thorough objective examination of the knee, during which various clinical tests are performed to evaluate potential joint deformities, objective instability, and meniscal injuries. The obtained score determines an objective evaluation grade codified using Roman letters. According to this scale, grade "A" is assigned to a knee with "normal, healthy" functionality, grade "B" is assigned to a knee with "nearly normal" functionality, grade "C" is assigned to a knee with "moderately abnormal" functionality, and grade "D" is assigned to a knee with "severely abnormal" functionality.
VAS (visual analog scale) | 24 months after surgery
  It is a unidimensional quantitative numeric pain rating scale with 10 points. The scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that specific moment. 0 means no pain and 10 indicates the worst possible pain.
SF-36 (Short Form-36 Health Survey) | 24 months after surgery
  It is the most well-known and widely used health-related quality of life measurement tool in international literature. It assesses various health concepts through 36 multiple-choice questions, with the data aggregated into 8 scales that investigate: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Additionally, there is one question about changes in health status over the past year.
Tegner Score | 24 months after surgery
  It allows for the estimation of a subject's level of physical activity with a score ranging from 0 to 10, where 0 represents 'incapacity' and 10 represents 'participation in competitive sports, such as national or international level soccer.' This score is the most commonly used to define the level of physical activity in patients with knee disorders. Additionally, the patient will be asked how many years they have been active in sports and whether the reason for reducing or ceasing activity is related to knee pathology or not.
Hip circonference | 24 months after surgery
  Measuring the thigh circumference at 5 cm and 15 cm above the superior pole of the patella allows for the assessment of muscle trophism in the subjects under examination, thereby evaluating the potential influence of the technique used on the knee's extensor apparatus.
Anterior knee pain / pain during knee flexion | 24 months after surgery
  To specifically assess the symptoms of the femoropatellar joint, patients will be asked to answer these questions in a dichotomous manner (YES/NO).
Patient satisfaction | 24 months after surgery
  In order to assess the level of patient satisfaction, they will be asked to respond to the question "Are you satisfied with the surgical intervention?" Once again, the response will be dichotomous.
Radiographic evaluation | 24 months after surgery
  The study will collect clinical and imaging data from patients to assess the development of osteoarthritis and other radiographic anomalies. If patients lack radiological documentation according to the study protocol post-intervention, weight-bearing lower limb X-rays and lateral projection X-rays of the operated knee will be conducted to evaluate osteoarthritis severity using the Kellgren-Lawrence scale. This scale categorizes osteoarthritis into 5 grades based on joint space reduction and osteophyte presence. Additionally, computer-assisted quantitative analyses will be performed on radiographic images at the collaborating facility for precise measurement of pre- and post-operative joint angles.
Complications or subsequent interventions | 24 months after surgery
  Any complications and subsequent interventions will be documented and recorded in the Case Report Form (CRF).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No